CLINICAL TRIAL: NCT02624245
Title: The Movement Control Training Associated With Conventional Physical Therapy is More Effective Than Conventional Physical Therapy Alone in Pain and Functional Performance?
Acronym: MCTACPTMECPTA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Paulo Roberto Garcia Lucareli, Professor, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: : PL004
Record Dates: First submitted 2015-12-02; First posted 2015-12-08 (Estimated); Last update posted 2015-12-08 (Estimated); Status verified 2015-12

CONDITIONS: Patellofemoral Pain Syndrome
MeSH Terms: conditions — Patellofemoral Pain Syndrome | interventions — Weight-Bearing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental: Conventional Physical Therapy (Experimental): Strength, this arm will receive hip and knee muscle strengthening with and without weight bearing.
  Interventions: Other: Conventional Physical Therapy
- Movement control training (Active Comparator): Movement control training, this arm will receive movement control training associated to muscle strengthening.
  Interventions: Other: Conventional Physical Therapy

INTERVENTIONS:
Other: Conventional Physical Therapy
  Other Names: hip abductors, lateral hip rotators and knee extensors strengthing exercises with and without weightbearing

SUMMARY:
Assess pain, performance function, hip and knee strength and kinematics of trunk and lower limbs during single leg hop test after movement control training associated to hip and knee muscle strengthening.

ELIGIBILITY:
Inclusion Criteria:

* Sedentary women,
* Previous knee pain last 3 months in at least two of the following activities: sitting for long periods, walk up or down stairs, squat, running and jumping

Exclusion Criteria:

* Lower limb surgery,
* Patella displacement
* Knee instability
* Heart or locomotor disorders which might influence the evaluation

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2013-05; Primary Completion 2014-08 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Pain | 4 weeks
  NRPS Score
Functional Performance | 4 weeks
  Single leg hop test distance

SECONDARY OUTCOMES:
Strength of hip and knee extensor muscles measured through hand-held dynamometer | 4 weeks
3D kinematic range of motion of hip adduction during single leg hop test | 4 weeks
3D kinematic maximum angular value of hip adduction during single leg hop test | 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Nove de Julho, São Paulo, São Paulo, Brazil